CLINICAL TRIAL: NCT03361475
Title: Community-based Mental Wellness Project for Adolescents and Adults SME (Sharing, Mind & Enjoyment) App - A Pilot Project
Brief Title: SME(Sharing, Mind & Enjoyment) App for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Dr Sun Yuying, Principle investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPH-MHP-TWGH01
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Mental Health Wellness 1
Keywords: Sharing; Mind; Enjoyment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention school (Experimental): One school workshop and a small talk were conducted first at the beginning of the programme, which was to promote SME and introduce the function of SME App for students, followed by downloading and using immediately to connect family members, then let them continue to use for one month with system reminder.
  Interventions: Behavioral: SME App
- Waitlist control schools (No Intervention): The intervention won't be provided during evaluation period and will be provided after the evaluation period

INTERVENTIONS:
Behavioral: SME App — The features in the App could be used in the future by linking with some platforms / existing services so that more SME messages can be sent to the students for sharing. One school workshop will be held to promote SME and introduce the function of SME App for students to download and use immediately to connect family members.
  SME App promotes SME via:
  * Express gratitude to family members (sharing)
  * Deliver positive messages regularly (mind)
  * Record physical and other joyful activities (enjoyment)
  * Increase knowledge and understanding of adolescent mental health problem (in particular the anxiety disorders)
  Arms: Intervention school

SUMMARY:
SME (Sharing, Mind, Enjoyment) App, A Pilot Project is part of the Community-based Mental Wellness Project for Adolescents and Adults, which aims at promoting sharing, mind and enjoyment and enhancing mental wellbeing. The Mental Wellness Project is financially supported by the Health Care and Promotion Fund from Food and Health Bureau and led by the School of Public Health, University of Hong Kong (HKU). This project primarily aims to promote the SME related behaviors of adolescents through the App. The evaluation will be conducted during the programme implementation stage. The effectiveness of the intervention, as well as the level of participation and ratings for the intervention, will be evaluated.

DETAILED DESCRIPTION:
A cluster randomized controlled trial design was adopted. The major subjects of SME (Sharing, Mind, Enjoyment) App Pilot Project RCT Study are 300-500 middle school students. Two schools will be recruited and randomized to each group. Schools will either be assigned to app intervention group or waitlist control group. The students in the intervention group will use the App for one month. Daily and Weekly tasks related to SME will be assigned through the App, and information related to mental health will be provided. The waitlist control group will be able to use the App after we finish all the assessments.

There will then be 4 assessments (pre-intervention, immediate post-intervention, one month and three months after) to evaluate the effects of the intervention programme. In the assessments, students will be asked to complete a questionnaire to measure the changes in SME (sharing, mind and enjoyment) related behaviors, changes of knowledge and attitude towards the anxiety disorder, changes of happiness and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Students (major subjects) (intervention group and control group):

  1. Chinese speaking
  2. Intact verbal and hearing abilities for interpersonal communication
  3. Reading and writing abilities for questionnaire completion
  4. Can use the smartphone
  5. Form 1 to 4 students
* Parents (intervention group):

  1. Chinese speaking
  2. Intact verbal and hearing abilities for interpersonal communication
  3. Reading and writing abilities for questionnaire completion
  4. Can use the smartphone
  5. With at least one child between form 1 to 4
* School principals/teachers/community partners (intervention group):

  1. Principals/teachers of intervention school or staffs of Tung Wah Group of Hospitals in partnership with HKU research team, who organize plan or implement the project
  2. Adults aged 18 or above
  3. Chinese speaking
  4. Intact verbal and hearing abilities for interpersonal communication
  5. Reading and writing abilities for questionnaire/individual in-depth interviews completion

Exclusion Criteria:

* Students who cannot read Chinese

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in the concept of Sharing, Mind and Enjoyment (SME) for adolescents and their family members. | T1: before the SME App workshop (baseline); T3: 1-month after baseline; T4: 3-month after baseline
  The outcome-based questionnaire will be used to evaluate participants' frequency of performing the suggested Sharing, Mind and Enjoyment (SME) related behaviours from baseline to three-month after baseline.

SECONDARY OUTCOMES:
Changes in the knowledge and understanding about mental health for adolescents and their family members. | T1: before the SME App workshop (baseline); T2: immediately after the SME App workshop ( post intervention ); T3: 1-month after baseline; T4: 3-month after baseline
  The outcome-based questionnaire will be used to evaluate participants' knowledge and understanding about anxiety disorder from baseline to three-month after baseline.
Changes in personal happiness from baseline to three-month after baseline | T1: before the SME App workshop (baseline); T3: 1-month after baseline; T4: 3-month after baseline
  Personal happiness will be assessed by Subjective Happiness Scale (SHS). SHS was rated on 7-point scale with 1 indicating not happiness at all and 7 indicating extreme happiness. To score the scale, the 4th item will be coded reversely and mean of the 4 items will be computed.
Changes in mental well-being from baseline to three-month after baseline | T1: before the SME App workshop (baseline); T3: 1-month after baseline; T4: 3-month after baseline
  Mental well-being will be assessed by validated Chinese version of 7-item Warwick Edinburgh Well-being Scale. Each item ranges from 1 to 5 and the scale will be scored by first summing the score for each of the 7 items and then transforming the total score for each person according to a conversion table.
Changes in individual and family health from baseline to three-month after baseline | T1: before the SME App workshop (baseline); T3: 1-month after baseline; T4: 3-month after baseline
  Self-perceived health, happiness and harmony at the individual and family level will be assessed by a 0-10 score at 3 time points
Satisfaction toward SME App Project | T2: immediately after the SME App workshop ( post intervention ); T3: 1-month after baseline; T4: 3-month after baseline
  Satisfaction towards the workshop, short interactive talk on SME and SME app will be assessed by programme evaluation measure
The social impact of the community-based engagement project | T4: 3-month after baseline
  The social impact of the community-based engagement project will be The satisfaction, ratings and opinions on SME App programme of school principal/teacher/community partner in the intervention group will be assessed qualitatively (individual in-depth interviews)
The process of community based intervention programme | up to 3 months
  The process evaluation on-site observation questionnaire will be used to assess the process of the community-based intervention programs.

CONTACTS AND LOCATIONS:
Overall Officials: Yuying Sun, Dr., Principal Investigator — Post-doctoral Fellow
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Sun Y, Wang MP, Ho SY, Chan CS, Man PKW, Kwok T, Wan ANT, Lam TH. A Smartphone App for Promoting Mental Well-being and Awareness of Anxious Symptoms in Adolescents: A Pilot Cluster Randomized Controlled Trial. Games Health J. 2022 Oct 3. doi: 10.1089/g4h.2021.0215. Online ahead of print. PMID 36194074